CLINICAL TRIAL: NCT04946760
Title: Effects of OMT on Gait Kinematics and Postural Control in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Kendi Hensel, DO, PhD, Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #2016-097
Record Dates: First submitted 2021-06-15; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease
Keywords: Osteopathic Manipulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Protocol (Sham Comparator): The sham protocol will consist of examination of the subject's active and passive range of motion in the spine and extremities, in the joints that would have been treated with OMT. The subject will be positioned in sitting, supine and lateral recumbent in a similar manner to that of the OMT group, but without providing an active intervention. To provide a sham for the OMT-WB protocol, subjects will lie supine with the physician's hands under the occiput, palms toward the table, so that the subject's head rests on the dorsal aspect of the physician's hands. The time used in the sham procedures will be approximately 20-25 minutes.
  Interventions: Other: Sham Manipulation
- Whole-Body Protocol (Experimental): The whole-body protocol will include all the techniques in the OMT-ND protocol, but will also include techniques focused on the expected cranial dysfunctions [Rivera-Martinez 2002]. The OMT-WB protocol will last approximately 25-30 minutes.
  The techniques will include:
  * Evaluation for strain pattern(s)
  * Occipitolatlantal decompression
  * Sphenobasilar synchondrosis decompression
  * Occipitomastoid suture V-spread
  * Temporal bone balancing
  * Venous sinus drainage technique
  Interventions: Other: Sham Manipulation
- Neck-down protocol (Experimental): The neck-down protocol takes into consideration previous relevant studies [Lopez 2011, Wells 1999]. OMT will be used bilaterally on the following areas with one or more techniques, including myofascial release, articulatory, muscle energy, and balanced ligamentous tension. The OMT-ND protocol will last approximately 15-20 minutes.
  * Cervical spine
  * Thoracic spine
  * Lumbar spine
  * Shoulder girdle
  * Sacroiliac joint
  * Innominates
  * Leg muscles (including psoas, piriformis, hamstring, adductors)
  * Ankles
  Interventions: Other: Sham Manipulation

INTERVENTIONS:
Other: Sham Manipulation — The sham protocol will consist of examination of the subject's active and passive range of motion in the spine and extremities, in the joints that would have been treated with OMT. The subject will be positioned in sitting, supine and lateral recumbent in a similar manner to that of the OMT group, but without providing an active intervention.

SUMMARY:
Parkinson Disease is a degenerative process that affects millions each year, and has devastating effects on patients and their families. The mobility symptoms that manifest as the disease progresses can result in social isolation as patients may be embarrassed or fear falling in public. One of the common risks resulting from the PD is falls. Falling in PD is primarily related to musculoskeletal issues such as muscular rigidity, postural instability & stooped posture. These kinds of manifestations should be amenable to treatment with OMT. There are studies showing the positive impact that OMT has on gait in PD, and a study showing improvement in balance in non-PD subjects. This investigation is designed to address these components via the following specific aims:

1. Identify the effects of a Neck-down OMT (OMT-ND) protocol on gait kinematics and postural control in Parkinson disease The investigators hypothesize that the application of an OMT protocol will improve gait kinematics and increase subjects' ability to respond to a postural challenge. The theoretical mechanism for this is due to the improved joint flexibility, improved proprioception and decreased muscle co-activation.
2. Determine the efficacy of Whole-body OMT (OMT-WB) protocol including cranial manipulation on gait kinematics and postural control in Parkinson disease The investigators hypothesize that the addition of a cranial manipulation protocol will further improve gait kinematics and increase subjects' ability to respond to a postural challenge. The theoretical mechanism for this is due to the improved arterial blood flow to the brain, which results from improving the cranial bone motion, maximizing venous drainage, and reducing any restrictions around the vestibular system.

DETAILED DESCRIPTION:
Disordered health does not simply progress in one direction from disease process, to disability, to handicap; rather, the process is a complex interaction between health conditions, body structure and function, environmental and personal factors, and limitations in activity and participation. Biologic,behavioral, environmental, and socioeconomic risk factors can all contribute to this progression. In the case of Parkinson disease (PD), this progression includes the degradation of balance and stability resulting in falls. Parkinson disease (PD) is the second most common neurodegenerative disease worldwide. It results from a lack of dopamine production within the substantia nigra, and is characterized by slowness of movement (bradykinesia), muscle rigidity (akinesia), postural instability, and resting tremor. As a result, PD patients have a characteristic short shuffling gait, with a loss of associated arm motion. Gait initiation is difficult and sudden freezing may impair components of movement such as turning. Postural instability and gait difficulty increase over the course of the disease, and expose PD patients to a nine times greater risk of falls. Falls can cause physical injuries such as fractures and/or head injuries leading to functional incapacity, increased risk of nursing home admission and higher mortality rate. Musculoskeletal manifestations of PD may be as impactful as the nervous system manifestations. For example, muscle rigidity associated with dopaminergic loss can lead to somatic dysfunction, which can impact posture and gait. Osteopathic medicine, with its philosophical understanding of the central role of the musculoskeletal system, is in an ideal model for this direction of research. Recent evidence has demonstrated OMT's efficacy in improving postural control in healthy older subjects. Wells et al., were the first to examine the effects of an OMT protocol in a cohort of persons with PD. While this study demonstrated a positive effect on gait kinematics, it investigation failed to examine static components of postural control, which are the most common cause of falls in PD.

The investigators have carefully designed this study to identify the effects that an OMT protocol has on gait kinematics and postural control in subjects with PD. This design compares the effectiveness of two OMT protocols: the Neck-Down (OMT-ND) protocol focuses on addressing biomechanical dysfunctions from the neck down; and the Whole-Body (OMT-WB) protocol, includes the ND techniques and adds specific Osteopathic Cranial Manipulative Medicine (OCMM) techniques to address dysfunctions in the head.

The investigators hypothesize that the application of an OMT protocol will improve gait kinematics and increase subjects' ability to respond to a postural challenge due to improved joint flexibility, improved proprioception and decreased muscle coactivation. The investigators hypothesize that the addition of a cranial manipulation protocol will further improve gait kinematics and increase subjects' ability to respond to a postural challenge. The theoretical mechanism for this is due to the improved arterial blood flow to the brain, which results from improving the cranial bone motion, maximizing venous drainage, and reducing any restrictions around the vestibular system.

The investigators also include a sham group to strengthen the internal validity of the OMT- ND and OMT-WB protocols. Research on OMT's specific effects is sometimes difficult to differentiate from placebo effects. Distinct placebo components include assessment and observation, therapeutic ritual, and a supportive patient-practitioner relationship. The sham treatment will control for these components with minimal impact on the biomechanical dysfunctions in our subjects.

The investigators plan to investigate the effect of these OMT protocols via the following specific aims:

1. Identify the effects of a Neck-down OMT protocol (OMT-ND) on gait kinematics and postural control in Parkinson disease;
2. Determine the efficacy of a Whole-body OMT protocol (OMT-WB) including cranial manipulation on gait kinematics and postural control in Parkinson disease.

The investigators' long-term goal is create a reproducible protocol that improves gait and postural control, and helps to reduce falls and improve quality of life in persons with PD. If the results validate the previous studies and prove the hypotheses, this study will advance osteopathic medicine by demonstrating OMT as a useful adjunct treatment in patients with PD. The investigators' expectation is that by improving gait and postural control, OMT can help PD patients reduce falls, which may allow them to be more active and lead a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* For PD participants: Neurologist-diagnosed idiopathic PD, H&Y stages 1.0-3.0
* Ability to stand independently for 1 minute and ambulate 100 yards independently
* Healthy (not under ongoing medical care for health problems that could impact performance on study tasks)
* for controls: age-matched healthy adults

Exclusion Criteria:

* Idiopathic PD in Hoehn & Yahr stages >3.0
* Previous surgical management of PD (pallidotomy, deep brain stimulation
* Central or peripheral nervous system disorders other than PD including, but not limited to multiple sclerosis, cerebral palsy, Alzheimer's diseases, or chronic fatigue syndrome
* Cognitive impairment as defined by the Mini-Mental Status Examination (<26 for subjects with PD and <24 for control subjects)
* Unable to stand independently for 1 minute and to walk independently for 100 yards
* Body weight >400lbs

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Timed up and Go test | Pre and immediately post intervention, change will be reported
  The "Timed Up and Go" Test (TUG), which measures the ability of participants to perform sequential mobility tasks that incorporate walking and turning. Specifically, in this timed test, participants begin in a seated position in an armchair. They are asked to rise, go forward 3m, turn around and sit back down. In older adults at risk for falls and persons with PD, the TUG has been found to possess excellent intra-tester reliability (0.94-0.96) and predictive validity, with increased times on the TUG relating to higher fall-risk.
Functional Reach Test | Pre and immediately post intervention, change will be reported
  The functional reach test (FR) is a simple balance task that tests the ability of a person to move their center of mass to the anterior limits of their base of support by measuring the distance a participant can reach forward from a quiet stance position. [Duncan, 1990; Duncan, 1992] The FR distance has previously been demonstrated to be predictive of fall risk in elderly persons, possess excellent test-retest reliability,[Brusse, 2005; Steffen, 2005] and can distinguish between those persons with PD with a history of falls from those with no falling history.

SECONDARY OUTCOMES:
Gait kinematics | Pre and immediately post intervention, change will be reported
  Kinetic, kinematic, and spatiotemporal measures will be gathered during gait using the predetermined comfortable walking speed. This will include joint angles, center of mass, center of pressure, stride length and stride width.
Postural control | Pre and immediately post intervention, change will be reported
  The postural control task in this investigation will also be assessed using the CAREN system by inducing perturbations on a dual-belt treadmill. Unexpected perturbations will be delivered in the forward and backward direction during static stance and straight-line ambulation by manipulating the speed and acceleration of the treadmill. Five perturbations will be delivered per direction (forward/backward), for a total of 10 perturbations per participant. Measure of body sway and time to stability will be collected.
  Outcome measures will be assessed using a 12-camera Motion Analysis system (Cortex Motion Analysis, Santa Rosa, CA).

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No